CLINICAL TRIAL: NCT00640419
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2 Study of the Safety and Efficacy of 0.7 mg/kg/Day and 1.4 mg/kg/Day of ABT-089 in the Treatment of Children With Attention Deficit-Hyperactivity Disorder (ADHD)
Brief Title: Safety and Tolerability Study of ABT-089 in Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-345
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — pozanicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: ABT-089
- 2 (Experimental)
  Interventions: Drug: ABT-089
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ABT-089 — Subjects will take 10 mg capsules and/or 40 mg tablets (actual dose based on weight) once daily for 6 weeks.
  Arms: 1; 2
Drug: placebo — Subjects will take placebo capsules and/or tablets (number of capsules or tablets will be based upon weight) once daily for duration of the study.
  Arms: 3

SUMMARY:
The purpose of this study is to test if the investigational medication ABT-089 is a safe and effective treatment for children with Attention Deficit Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily signed an informed consent form.
* Meet diagnostic criteria for attention-deficit/hyperactivity disorder (ADHD) based on detailed evaluation and interview with parent(s).
* Subject is generally in good health based on medical history, physical examination, clinical lab tests and ECG.
* Subject weights at least 37 pounds (17 kg)
* Female subjects of child-bearing potential must have a negative urine pregnancy test at screening and baseline and agree to comply with applicable contraceptive requirements.
* Subject can swallow pills and subjects and parents are able to keep required appointments for clinic visits and all tests, including blood draws and examinations.

Exclusion Criteria:

* Subject has a current or past diagnosis of bipolar disorder, psychosis, autism, Asperger syndrome, pervasive developmental disorder, tics, Tourette syndrome, mental retardation, seizure disorder or traumatic brain injury.
* Current diagnosis of obsessive-compulsive disorder, eating disorder, anxiety disorder or depressive disorder requiring treatment of any kind.
* Subject has a history of, or ongoing, serious medical problem.
* Subject has a history of significant allergic reaction to any drug.
* Subject is planning to begin any type of behavioral or psychotherapy for treatment of ADHD.
* Subject requires ongoing treatment with any psychiatric medication.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
ADHD-RS-IV (HV) | Screening, Day -1, Day 7, Day 14, Day 28, Day 42

SECONDARY OUTCOMES:
CSHQ | Day-1, Day 28, Day 42
CGI-P | Day -1, Day 21, Day 42
BRIEF | Day -1, Day 28, Day 42
CGI-ADHD-S | Screening, Day -1, Day 7, Day 14, Day 28 and Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Laura Gault, Study Director — AbbVie
Locations (13):
- United States (13):
  - Site Reference ID/Investigator# 7536, Little Rock, Arkansas
  - Site Reference ID/Investigator# 7954, Bradenton, Florida
  - Site Reference ID/Investigator# 7543, Jacksonville, Florida
  - Site Reference ID/Investigator# 7542, Orlando, Florida
  - Site Reference ID/Investigator# 7537, Libertyville, Illinois
  - Site Reference ID/Investigator# 7561, Overland Park, Kansas
  - Site Reference ID/Investigator# 7560, Troy, Michigan
  - Site Reference ID/Investigator# 7559, Omaha, Nebraska
  - Site Reference ID/Investigator# 7541, Las Vegas, Nevada
  - Site Reference ID/Investigator# 7564, Oklahoma City, Oklahoma
  - Site Reference ID/Investigator# 7538, Portland, Oregon
  - Site Reference ID/Investigator# 7540, Memphis, Tennessee
  - Site Reference ID/Investigator# 7544, Bellevue, Washington

REFERENCES:
- [Derived] Wilens TE, Gault LM, Childress A, Kratochvil CJ, Bensman L, Hall CM, Olson E, Robieson WZ, Garimella TS, Abi-Saab WM, Apostol G, Saltarelli MD. Safety and efficacy of ABT-089 in pediatric attention-deficit/hyperactivity disorder: results from two randomized placebo-controlled clinical trials. J Am Acad Child Adolesc Psychiatry. 2011 Jan;50(1):73-84.e1. doi: 10.1016/j.jaac.2010.10.001. Epub 2010 Nov 25. PMID 21156272